CLINICAL TRIAL: NCT03469752
Title: Latino Fathers Promoting Healthy Youth Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-68001-24921
Record Dates: First submitted 2018-03-08; First posted 2018-03-19 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Diet Modification; Physical Activity; Parenting; Adolescent Obesity
Keywords: Hispanic Latino families
MeSH Terms: conditions — Motor Activity; Pediatric Obesity | interventions — Prenatal Education

STUDY DESIGN:
Intervention Model Description: Randomized-controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 8 weekly education sessions 2.5 hours
  Interventions: Behavioral: Parent education classes
- Wait-list control group (No Intervention): No education sessions

INTERVENTIONS:
Behavioral: Parent education classes — 8 weekly classes for fathers and youth (10-14 years) at community centers focused on improving parenting skills, youth energy balance related behaviors and weight status
  Arms: Intervention group

SUMMARY:
The purpose of this study is to evaluate the efficacy of Latino parent-focused education that combines enhancing parent engagement, building quality parent-child relationships, promoting healthy eating and physical activity, and engaging families with community resources for healthy foods on youth energy balance related behaviors and weight status.

DETAILED DESCRIPTION:
The Latino Parents Promoting Healthy Youth Behavior Project aims to develop and evaluate the effectiveness of an intervention to prevent obesity among Latino youth (10-14 yrs) by engaging parents and their families in culturally and linguistically appropriate education. The goal of this project is to prevent overweight and obesity in Latino adolescents by increasing the frequency of positive paternal or maternal (or other caregiver) parenting practices related to the food and physical activity environment in the home (role modeling, availability, expectations, communication) which will improve weight status of children by improving energy balance related behaviors (EBRBs) - eating fruits and vegetables and limiting soft drink, sweets, salty snacks, and fast food consumption, limiting screen time and increasing physical activity).

Objective 1) To adapt, implement and evaluate efficacy of a curriculum specifically for Latino families, using Community-Based Participatory Research (CBPR) that incorporates parenting education to increase frequency of parenting practices (role modeling, availability, expectations, communication) to improve EBRBs and weight status of youth.

Objective 2) To evaluate the efficacy of Latino parent-focused education that combines enhancing parent engagement, building quality parent-child relationships, promoting healthy eating and physical activity, and engaging families with community resources for healthy foods on youth EBRBs and weight status.

Formative research and planning will be completed in Years 1-2 including focus group interviews and consultation with community partners and a Parent Advisory Board. An existing 8-session course curriculum will be adapted. The adapted curriculum will be pilot-tested with a small group of parents and children in a single group, pre-post design, and revised as needed.

In years 2 to 4, a randomized-controlled trial (RCT) will be conducted based on full implementation of the adapted curriculum by collaborating agencies with the support of U of MN Extension. Training will be designed and implemented among community partner and U of MN Extension staff who will be implementing the program at local sites.

The RCT will be implemented at two organizations in each of years 2, 3 and 4 in a staggered fashion. In year 5, data will be analyzed, reports developed, papers written and submitted for publication, and results will be reported back to community collaborators (organizations and individuals).

Hypothesis:

1. Compared to a delayed-treatment control group at immediate post-course and 3 months post-course, statistically significant changes will be observed in the home food and physical activity environment and frequency of related paternal and maternal parenting practices (making fruits, vegetables, and opportunities for physical activity more available and sugar-sweetened beverages (SSBs), sweets, salty snacks, fast food and opportunities for sedentary behaviors less available; role modeling of positive EBRBs, setting expectations and rules related to improvements in EBRBs, and increased frequency of parent-youth communication regarding youth EBRBs).
2. Compared to a delayed-treatment control group at immediate post-course and 3 months post-course, youth in the treatment group will have statistically significant improvements in EBRBs including increased fruit and vegetable intake, increased physical activity, lower intake of SSBs, sweets, salty snacks and fast food, decreased screen time/sedentary time, and stable weight status.

ELIGIBILITY:
Inclusion Criteria:

* Latino adolescent 10-14 years

Exclusion Criteria:

* Not identifying as a Latino adolescent 10-14 years

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
3 24-hour diet recalls | Baseline to 3 months
  Dietary intake (fruits, vegetables, sweetened beverages, sweets and salty snacks, family meals)
Physical activity | Baseline to 3 months
  Physical activity survey

SECONDARY OUTCOMES:
Parenting practice survey | Baseline to 3 months
  Frequency of role modeling, setting expectations, making opportunities for healthy choices available

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baltaci A, Hurtado Choque GA, Davey C, Reyes Peralta A, Alvarez de Davila S, Zhang Y, Gold A, Larson N, Reicks M. Padres Preparados, Jovenes Saludables: intervention impact of a randomized controlled trial on Latino father and adolescent energy balance-related behaviors. BMC Public Health. 2022 Oct 18;22(1):1932. doi: 10.1186/s12889-022-14284-5. PMID 36258168